CLINICAL TRIAL: NCT06332612
Title: Repurposing Metformin for the Treatment of Oral Submucous Fibrosis: Unraveling Novel Signaling Pathways In Vitro and Advancing to Clinical Trial"
Brief Title: Metformin Repurposing in Oral Submucous Fibrosis: Unveiling In Vitro Signaling Pathways, Progressing to Clinical Trial
Acronym: MROSF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr. Afifa Razi, Professor, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8420224AROM
Record Dates: First submitted 2024-02-22; First posted 2024-03-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Oral Submucous Fibrosis
Keywords: Oral Submucous Fibrosis; Metformin; Randomized Controlled Clinial Trial; TGF Beta; Smad2/ 3 Signaling; Wnt Signaling
MeSH Terms: conditions — Oral Submucous Fibrosis; Camurati-Engelmann Syndrome | interventions — Metformin; betamethasone-17,21-dipropionate; Betamethasone Valerate; Pentoxifylline

STUDY DESIGN:
Intervention Model Description: 1. In Vitro (Cell Line) Study Design: Experimental in vitro study using OSF cell lines.
  Groups:
  * Metformin-treated
  * Control (untreated)
  * Vehicle control Clinical Trial Study Design: A pilot Randomized Controlled Trial (RCT) translating the in vitro findings into a clinical setting. It would be a single-blind, placebo-controlled designAll groups will undergo a 24-week intervention phase. Group 1 will receive standard treatment including topical cream betamethasone thrice daily and Pentoxifylline tablet 400 mg twice daily. Group 2 will receive Metformin 500 mg thrice daily. Group 3 will receive topical cream metformin thrice daily. All groups will be instructed to perform a stick mouth opening exercise twice daily, alternating sides, holding the stick for 10 minutes on each side, with a 10-minute rest in between. All groups will be single blinded to the intervention.
Who Masked: Participant
Masking Description: It would be a single-blind, placebo-controlled design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard (Active Comparator): Group 1: Standard treatment with topical cream betamethasone and Pentoxifylline tablet.
  Interventions: Drug: betamethasone dipropionate; Drug: Pentoxifylline
- MetforminO (Experimental): Metformin 500 mg thrice daily.
  Interventions: Drug: Metformin Hydrochloride
- MetforminT (Experimental): Topical cream metformin thrice daily
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Group B will receive Metformin 500 mg thrice daily. Group C will receive topical cream metformin thrice daily.
  Other Names: Glucophage
  Arms: MetforminO; MetforminT
Drug: betamethasone dipropionate — Group 1will recieve topical cream betamethasone thrice daily
  Other Names: Betnovate
  Arms: Standard
Drug: Pentoxifylline — Group 1 will receive Pentoxifylline tablet 400 mg twice daily
  Other Names: Trental
  Arms: Standard

SUMMARY:
OSF is a widespread health issue in Asian countries, notably Pakistan, linked to the consumption of pan, chalia, and gutka, affecting a rising number of young individuals as an epidemic. This condition significantly impairs oral function, resulting in ulcers and chronic lesions, often progressing to oral cancer. Current treatments focus on symptom relief and halting disease progression. This study explores the repurposing of metformin, an FDA-approved drug with antifibrotic properties, for OSF treatment. Our objective is to unveil its therapeutic potential and comprehend its impact on the dysregulated signaling pathways associated with OSF. This research offers promising insights for an enhanced management approach, providing hope for those grappling with this debilitating condition

DETAILED DESCRIPTION:
OSF stands as a persistent inflammatory and potentially malignant condition affecting the oral cavity, marked by progressive fibrosis of the oral mucosa. The spectrum of its manifestations spans from initial inflammation to the gradual emergence of fibrous bands, leading to restricted mouth opening and mucosal rigidity. Common symptoms encompass burning sensations, difficulty in swallowing, and alterations in taste perception. This health concern has gained prominence in Pakistan, experiencing a worrisome surge in prevalence from 8.3/105 to 16.2/105 in recent years. Formerly confined to Southeast Asia, OSF has now transcended borders, manifesting in Asian immigrant communities in Britain and America, evolving into a global oral potential malignant disorder (OPMD) with a malignant rate of 9.13% .

Presently, the corticosteroid-based approach effectively reduces inflammation in OSF but falls short in addressing the underlying molecular mechanisms contributing to fibrosis. Furthermore, the prolonged use of corticosteroids raises concerns about adverse effects, including mucosal atrophy and compromised tissue integrity. This study aims to investigate the potential of metformin, a recognized emerging drug for treating fibrosis, and its anti-fibrotic properties in various organs. The established safety profile of metformin adds an advantageous aspect to its potential applications.

Numerous studies indicate that metformin exhibits anti-fibrotic effects by inhibiting TGF-β1 production, reducing phosphorylation and nuclear translocation of Smad2/3. Additionally, metformin inhibits Smad2/3 phosphorylation independently and activates AMPK, hindering Smad3 phosphorylation. The impact on reactive oxygen species (ROS) generation moderates TGF-β1-induced Smad2/3 phosphorylation and myofibroblast differentiation.Metformin has shown promise in hindering collagen production and promoting trans differentiation in various organ, including the lung, kidney, heart and adipose tissue. A clinical trial reported metformin therapy's impact on postmenopausal ovaries, patients with type 2 diabetes mellitus (T2DM) exhibited isotropic collagen organization and reduced fibrosis during oophorectomy.The observed risk reduction for ovarian cancer in T2DM women using metformin suggests its potential as an ovarian cancer prophylaxis. Despite conflicting clinical trial results in liver fibrosis, metformin consistently improves hepatocyte damage and inflammation. Clinical trials have explored the role of metformin antitumor activity when combined with conventional chemotherapeutic drugs and in idiopathic pulmonary fibrosis it inhibits TGFβ1, suppressing collagen formation, activating PPARγ signaling and inducing lipogenic differentiation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with OSF- palpable bands on oral examination
2. Patients with limited mouth opening due to OSF
3. Patients who have not received any treatment for OSF in the previous three months
4. Patients with habits of pan, Chalia, Ghutka
5. Age group between 18 and 45 years

Exclusion Criteria:

1. Patients presenting with both OSCC and OSF
2. Patients with limited mouth opening due to impaction of the third molar (impaction of third molar results in limited mouth opening hence such patients are excluded since limited mouth opening due to third molar impaction can be mistaken for OSF).
3. Patients with limited mouth opening due to temporomandibular joint disorder (temporomandibular joint disorders can limit the ability of patient to open their mouth and hence can be mistaken for OSF)
4. Any history of Metformin intolerance or contraindications.
5. Presence of other severe medical conditions along with drug therapy.
6. Pregnancy or lactation.
7. Participation in other clinical trials concurrently.
8. Inability to provide informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Cell Viability | 8 months
  Cell Viability by MTT Assay Unit: Percentage Assessment of cell viability will be reported as a percentage of untreated control cells.
Cytotoxicity | 8 Months
  Cytotoxicity Unit: Percentage Measurement of cytotoxicity will be presented as a percentage relative to untreated control cells.
Morphological Changes Cell Shape | 8months
  Unit: Qualitative description Cell shape alterations will be described qualitatively based on microscopic observations.
Morphological Change Cell Density | 8 months
  Unit: Cells per unit area Changes in cell density will be quantified and reported as cells per unit area. Sub-Measure 3: Extracellular Matrix (ECM) Structure Unit: Qualitative description Alterations in ECM structure will be qualitatively assessed.
Morphological Change Extracellular Matrix (ECM) Structure | 8 months
  Extracellular Matrix (ECM) Structure Unit: Qualitative description Alterations in ECM structure will be qualitatively assessed.
Cell Migration Assays | 8months
  Unit: Distance migrated (micrometers) The extent of cell migration will be quantified as the distance migrated from the original point.
Cell Invasion Assays | 8 months
  Unit: Invaded area (e.g., square millimeters) Assessment of cell invasion will be presented as the invaded area relative to untreated control cells.
Apoptosis Analysis | 8months
  Unit: Percentage Apoptotic cells will be quantified and reported as a percentage of the total cell population.
Assess Signaling pathway with optimal metformin concentration | 9 months
  To evaluate the effect of TGF-beta Smad 2/3 and wnt/b-catenin signaling pathways in vitro

SECONDARY OUTCOMES:
Clinical Oral Mucosal Characteristics | 9 months
  Unit: Descriptive score (based on a scale ranging from 0 to 3 (normal to severe).0=No changes 1=Soreness 2=Soreness and ulceration 3=Soreness, ulceration and ability to use a liquid diet only
Patient Burning sensation pain | 9 months
  Unit: Units on a scale (Verbal numeric rating scale graded on a 10-point scale from 0 to 10, where 0 indicated no burning sensation while 10 represented the worst burning sensation)
Patient Mouth Opening | 9 months
  Unit: Millimeters on a scale of Grade 0 = > 35 mm, Grade1= 26-35mm, Grade 2= 15-25mm, Grade 3: < 10mm

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The decision not to share Individual Participant Data (IPD) may be based on several considerations and could be influenced by institutional policies, ethical guidelines, and practical constraints.Sharing individual-level data may risk the identification of study participants, even with anonymization efforts, especially in smaller studies or specific populations

REFERENCES:
- [Result] Yang SF, Wang YH, Su NY, Yu HC, Wei CY, Yu CH, Chang YC. Changes in prevalence of precancerous oral submucous fibrosis from 1996 to 2013 in Taiwan: A nationwide population-based retrospective study. J Formos Med Assoc. 2018 Feb;117(2):147-152. doi: 10.1016/j.jfma.2017.01.012. Epub 2017 Apr 5. PMID 28390753
- [Result] Shen YW, Shih YH, Fuh LJ, Shieh TM. Oral Submucous Fibrosis: A Review on Biomarkers, Pathogenic Mechanisms, and Treatments. Int J Mol Sci. 2020 Sep 30;21(19):7231. doi: 10.3390/ijms21197231. PMID 33008091
- [Result] Septembre-Malaterre A, Boina C, Douanier A, Gasque P. Deciphering the Antifibrotic Property of Metformin. Cells. 2022 Dec 16;11(24):4090. doi: 10.3390/cells11244090. PMID 36552855
- [Result] Wu M, Xu H, Liu J, Tan X, Wan S, Guo M, Long Y, Xu Y. Metformin and Fibrosis: A Review of Existing Evidence and Mechanisms. J Diabetes Res. 2021 Apr 29;2021:6673525. doi: 10.1155/2021/6673525. eCollection 2021. PMID 34007848
- [Result] Teague TT, Payne SR, Kelly BT, Dempsey TM, McCoy RG, Sangaralingham LR, Limper AH. Evaluation for clinical benefit of metformin in patients with idiopathic pulmonary fibrosis and type 2 diabetes mellitus: a national claims-based cohort analysis. Respir Res. 2022 Apr 11;23(1):91. doi: 10.1186/s12931-022-02001-0. PMID 35410255
- [Result] Pimentel I, Lohmann AE, Ennis M, Dowling RJO, Cescon D, Elser C, Potvin KR, Haq R, Hamm C, Chang MC, Stambolic V, Goodwin PJ. A phase II randomized clinical trial of the effect of metformin versus placebo on progression-free survival in women with metastatic breast cancer receiving standard chemotherapy. Breast. 2019 Dec;48:17-23. doi: 10.1016/j.breast.2019.08.003. Epub 2019 Aug 22. PMID 31472446